CLINICAL TRIAL: NCT03798860
Title: Monitoring of Donor-specific Antibodies (DSA) After Combined Treatment with Immunoglobulin a and Immunoglobulin M-enriched Intravenous Human Immunoglobulins and Plasmapheresis and Rituximab in Lung Transplantation
Brief Title: Monitoring of Donor-specific Antibodies After Treatment with Immunoglobulins, Plasmapheresis and Rituximab in Lung Transplantation
Status: Recruiting | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: DSA-2018
Record Dates: First submitted 2018-09-26; First posted 2019-01-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Lung Transplantation; Donor-specific Anti-human Leukocyte Antigen(HLA) Antibodies
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: blood samples — For performing the Luminex solid phase assay (SPA) test, 7.5 ml of patient whole blood are collected from a peripheral vein.

SUMMARY:
Single-arm, prospective observational study

DETAILED DESCRIPTION:
This is an observational study to monitor the treatment of donor-specific antibodies in lung transplant recipients with detection of donor-specific antibodies. All consented subjects will be approached for participation. The study will evaluate the effectiveness of the treatment protocol of donor-specific antibodies with Immunoglobulins or combined treatment with Immunoglobulins, Plasmapheresis and Rituximab after lung transplantation.

ELIGIBILITY:
Inclusion Criteria:

* all patients after lung transplantation with detection of donor-specific antibodies

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients after lung transplantation with detection of donor-specific antibodies
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Donor-specific Antibodies Clearance | 6, 12, 18, 24 months
  The DSA clearance is defined as absence of DSA in the Luminex test, which is performed every 6 months after treatment end.

SECONDARY OUTCOMES:
Graft survival | 1, 3, 5 years
  Graft survival is defined as freedom from mortality and re-transplantation
Incidence of acute cellular and humoral rejections and chronic lung allograft dysfunction (CLAD) | 1, 3, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Ius, Dr., Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Department of Cardiothoracic, Transplant and Vascular Surgery, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No